CLINICAL TRIAL: NCT00605553
Title: A Randomized, Double-blind, Placebo Controlled, Two-way Cross-over Study to Explore the Effects of 7 Days of Dosing With SYN115 20 mg p.o. BID or 60 mg p.o. BID on Clinical and fMRI Response to Intravenous Levodopa in Patients With Mild to Moderate Parkinson's Disease
Brief Title: Study to Evaluate SYN115 in Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biotie Therapies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYN115-CL01
Record Dates: First submitted 2008-01-15; First posted 2008-01-31 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — tozadenant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Active medication Tozadenant 20 mg oral capsules with a daily dosage of either 20 mg BID or 60 mg BID
  Interventions: Drug: Tozadenant
- 2 (Placebo Comparator): Crossover from arm 1 to arm 2 with one week washout. One of the arms is placebo control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo oral capsules
  Placebo for 7 days
  Arms: 2
Drug: Tozadenant — 20 mg oral capsules with a daily dosage of either 20 mg BID or 60 mg BID
  Other Names: A2a antagonist; SYN115
  Arms: 1

SUMMARY:
This is an exploratory study to evaluate if SYN115 has an effect on Parkinson's disease as measured by clinical symptoms and brain images using magnetic resonance imaging (MRI) when a function test is administered.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, two-way crossover study in which each patient will act as their own control. Each patient enrolled will receive both SYN115 (20 mg or 60 mg) and placebo separated by a minimum of one week washout between periods. An adaptive design will be used to determine if SYN115 elicits effects relevant to PD in the fewest number of patients by performing interim analyses in successive cohorts of patients receiving 60 or 20 mg.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease
* Hoen and Yahr stage 1-3
* On stable dose of anti-parkinsons treatment for 30 days prior to screening
* Age 40 to 75 years
* Sign an IRB approved informed consent
* Men and women agree to use adequate birth control
* ECG measurements are within normal limits
* Able to understand study requirements

Exclusion Criteria:

* Secondary Parkinson's (drug induced or post stroke)
* Received treatment with other investigational drug 30 days prior to study entry
* Using disallowed medications
* Significant neurological illness other than Parkinson's
* IQ less than 70 on IQ test
* MMSE score < or = 23
* History of psychosis or on anti-psychotic medication
* Current serious medical illness
* History of substance abuse
* History of head injury with loss of consciousness
* History of brain surgery
* Contraindications to MRI like claustrophobia, metal implants or other implantable devices
* Abnormal liver function tests and/or hepatitis or cholangitis
* Gilberts disease
* Pregnant or nursing
* Known hypersensitivity to SYN115

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
This is an exploratory study to evaluate effects of SYN115 in patients with PD, as determined by clinical and fMRI evaluation. The results of this initial study will help determine the range to be used in subsequent studies. | Before treatment and at the end of each treatment period

SECONDARY OUTCOMES:
Pittsburgh side effect scale | Before, after the first dose and end of each treatment period
VAS for overall well being, dizziness/light-headedness, nausea/vomiting, mood anxiety | Before, after the first dose and end of each treatment period
Measurement of motor symptoms of Parkinson's disease and tapping speed | Before, after the first dose and end of each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Steve Bandak, MB BS MRCP, Study Chair — Synosia Therapeutics; Ann Neale, RN, Study Director — Synosia Therapeutics; Uwe Meya, MD, Study Chair — Synosia Therapeutics; Kevin J Black, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University St. Louis, St Louis, Missouri, United States

REFERENCES:
- [Result] Black KJ, Campbell MC, Dickerson W, Creech ML, Koller JM, Chung SC, Bandak SI: A randomized, double-blind, placebo-controlled cross-over trial of the adenosine 2a antagonist SYN115 in Parkinson disease. Neurology 74(9): A317, 2010.
- [Result] Black KJ, Koller JM, Campbell MC, Gusnard DA, Bandak SI. Quantification of indirect pathway inhibition by the adenosine A2a antagonist SYN115 in Parkinson disease. J Neurosci. 2010 Dec 1;30(48):16284-92. doi: 10.1523/JNEUROSCI.2590-10.2010. PMID 21123574